CLINICAL TRIAL: NCT01789528
Title: A Phase 1, Open-label, Multiple-dose, Single Centre Study to Investigate the Effect of Administration of CAZ-AVI and CXL on the Intestinal Flora of Healthy Volunteers.
Brief Title: A Study to Investigate the Effect of Administration of Ceftazidime-avibactam (CAZ-AVI) and Ceftaroline Fosamil -Avibactam (CXL) on the Intestinal Flora of Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D4280C00023
Record Dates: First submitted 2013-02-04; First posted 2013-02-12 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Pharmacokinetics; Open Label; CAZ-AVI; CXL; Effect on Intestinal Flora; Safety
Keywords: Phase I,; open label,; CAZ-AVI,; CXL,; healthy volunteers,; intestinal flora.
MeSH Terms: interventions — KPNA1 protein, human

ARMS (1):
- CAZ-AVI or CXL (Experimental): Cohort 1: CAZ-AVI (2000 mg ceftazidime and 500 mg avibactam) by intravenous infusion given over 2 hours, every 8 hours
  Cohort 2: CXL (600 mg ceftaroline fosamil and 600 mg avibactam)
  Interventions: Drug: CAZ-AVI; Drug: CXL

INTERVENTIONS:
Drug: CAZ-AVI — IV infusion
  Other Names: Cohort 1
Drug: CXL — IV infusion
  Other Names: Cohort 2

SUMMARY:
The purpose of this study is to investigate the effect of administration of CAZ-AVI and CXL on the intestinal flora of male and female healthy volunteers after multiple administrations over 7 days. An assessment of the effect on intestinal flora is an important aspect to understand for the safe clinical use of the investigational products and is expected by regulatory agencies.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures
2. Healthy male and female volunteers aged 18 to 45 years (inclusive) with suitable veins for cannulation or repeated venepuncture.

   Females: Female healthy volunteers are authorised to participate in this study if both of the following criteria are met:
   1. A negative serum pregnancy test BOTH at screening AND at admission to the study centre.
   2. Agrees not to attempt pregnancy while receiving investigational product and for a period of 7 days after last investigational product administration, and agrees to the use of acceptable methods of contraception (according to instructions) prior to, during, and for 7 days after the last investigational product administration.
3. Have a body mass index (BMI) between 19 and 30 kg/m2.

Exclusion Criteria:

1. History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
2. Any clinically significant abnormalities in physical examination, ECG, clinical chemistry, haematology, coagulation, or urinalysis results, as judged by the investigator.
3. Pregnant or breastfeeding female healthy volunteers.
4. History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the healthy volunteer at risk because of participation in the study, or influence the results or the healthy volunteer's ability to participate in the study.
5. Known history of Clostridium difficile infection in last 3 months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Changes in the intestinal flora of healthy subjects after administration of ceftazidime-avibactam (CAZ-AVI) and ceftaroline fosamil -avibactam (CXL). | Change from baseline (Day-1) at Day 2, 5, 7, 10, 14 and 21
  The number and types of microorganisms in faeces.

SECONDARY OUTCOMES:
Safety and tolerability | Screening up to 12 days after discharge from study site
  Adverse event, ECG, safety laboratory assessments, physical examinations and vital signs.
Pharmacokinetics of CAZ-AVI in healthy volunteers | Days 1, 2 and 5: Pre-dose and 2 hours post dose. Day 7: pre-dose, 0.5, 1, 1.5, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 6, 8, 12, and 24 hours post dose (Day 8)
  On Day 7, the following pharmacokinetic parameters will be calculated when applicable:
  Maximum plasma concentration (Cmax), time of Cmax (tmax), time of last quantifiable plasma concentration (last), area under the plasma concentration-time curve during the dosing interval (AUC(0-τ)), area under the plasma concentration time curve from zero to the time of the last quantifiable concentration (AUC(0-t)), half-life (t½), systemic plasma clearance (CL), apparent plasma clearance (CL/F), volume of distribution at steady state (Vss), and apparent volume of distribution (Vz/F).
Pharmacokinetics of CXL in healthy volunteers | Days 1, 2 and 5: Pre-dose and 1 hour post dose. Day 7: pre-dose, 0.5, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 5, 7, 8, 12, and 24 hours post dose (Day 8)
  On Day 7, the following pharmacokinetic parameters will be calculated when applicable:
  Maximum plasma concentration (Cmax), time of Cmax (tmax), time of last quantifiable plasma concentration (last), area under the plasma concentration-time curve during the dosing interval (AUC(0-τ)), area under the plasma concentration time curve from zero to the time of the last quantifiable concentration (AUC(0-t)), half-life (t½), systemic plasma clearance (CL), apparent plasma clearance (CL/F), volume of distribution at steady state (Vss), and apparent volume of distribution (Vz/F).
To measure CAZ-AVI and CXL plasma and faecal concentrations using bioactivity techniques. | Day -1, 2, 5, 7, 10, 14 and 21
  The concentrations of CAZ-AVI and CXL will be determined in plasma and faecal samples.
To describe the in vitro susceptibility of new colonizing bacteria of the intestinal microflora to CAZ-AVI and CXL during and after CAZ-AVI and CXL administration. | Day -1, 2, 5, 7, 10, 14 and 21
  Minimal inhibitory concentration (MIC) for CAZ-AVI and CXL will be determined for new colonizing bacteria from faecal samples.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Newell, MD, Study Director — AstraZeneca R&D, Alderly Park, Mereside, SK 104TG, Macclesfield, Cheshire, United Kingdom; Sandhia Ponnarambil, MD, Study Chair — AstraZeneca R&D Alderly Park, Parklands, SK 104TF, Macclesfield, Cheshire, United Kingdom; Georgios Panagiotidis, MD, Principal Investigator — Clinical Pharmacology Trial Unit, Karolinska University Hospital Huddinge, SE-141 86 Stockholm, Sweden
Locations (1):
- Research Site, Stockholm, Sweden